CLINICAL TRIAL: NCT05292560
Title: A Randomized Controlled Trial on the Effectiveness of a Positive Psychology App for Adults in the General Population Dealing With Negatives Consequences of the Corona Crisis
Brief Title: The Effectiveness of a Positive Psychology App in the General Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Twente (Other)
Responsible Party: Principal Investigator, Jannis Kraiss, Assistant Professor, University of Twente
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 220106
Record Dates: First submitted 2022-03-01; First posted 2022-03-23 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-11

CONDITIONS: Mental Health; Well-being; Depression; Anxiety; Adults; App; Positive Psychology
MeSH Terms: conditions — Psychological Well-Being; Depression; Anxiety Disorders; Alzheimer Disease

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Positive psychology app (Experimental)
  Interventions: Other: Training in positivity
- Waiting list (Other)
  Interventions: Other: Training in positivity

INTERVENTIONS:
Other: Training in positivity — The University of Twente developed an evidence-based positive psychology app that is aimed at increasing mental well-being and resilience (Training in positivity; TiP). TiP consists of a 3-week structured intervention, in which participants do two exercises every week for 6 days, aimed at increasing resilience and mental well-being. An exercise takes an average of 15 minutes per day.

SUMMARY:
The corona crisis has a negative impact on the mental wellbeing of the Dutch population. Positive psychology exercises (PPOs) can potentially improve mental well-being and reduce mild and moderate psychological complaints. Previous research has shown moderate to large effects of PPOs on well-being in people with reduced wellbeing and psychological symptoms at baseline. The University of Twente developed an app (Training in Positivity; TiP) based on an effective intervention. The goal of this study is to investigate the effectiveness of TiP in the general population in people experiencing reduced mental wellbeing as a result of the corona crisis. People using the app will be compared to a waiting list control group.

ELIGIBILITY:
Inclusion Criteria:

1. The participant is at least 18 years old
2. The participant has an e-mail address and is in possession of a smartphone or tablet with access to the internet.
3. The participant is willing to do a positive psychology exercise 6 days a week for 3 weeks
4. The participant has sufficient command of the Dutch language to be able to complete questionnaires and exercises.
5. The participant gives consent to participate in the study using the online informed consent procedure.

Exclusion Criteria:

1. The presence of severe anxiety symptoms: a score of 15 or higher on the Generalized Anxiety Disorder 7 items (GAD-7)
2. The presence of severe depressive symptoms: a score of 20 or higher on the Patient Health Questionnaire (PHQ-9).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2022-04-04 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
Mental well-being | Change from baseline mental well-being at 3 weeks (T1) and change from baseline mental well-being at 3 months (T2).
  Mental well-being measured with the 14-item Mental Health Continuum-Short Form. Scores are calculated as mean scores and can range from 0 to 5. Higher scores indicate more mental well-being.

SECONDARY OUTCOMES:
Ability to adapt | Change from baseline ability to adapt at 3 weeks (T1) and change from baseline mental well-being at 3 months (T2)
  Measured with the 10-item Generic sense of ability to adapt scale. Scores are calculated as sum scores and can range from 10 to 50. Higher scores indicate more ability to adapt.
General self-efficacy | Change from baseline general self-efficacy at 3 weeks (T1) and change from baseline mental well-being at 3 months (T2)
  Measured with the 10-item General Self-Efficacy Scale. Scores are calculated as sum scores and can range from 10 to 40. Higher scores indicate more general self-efficacy.
Savoring | Change from baseline savoring at 3 weeks (T1) and change from baseline mental well-being at 3 months (T2)
  Measured with the 24-item Savoring Beliefs inventory. Scores are calculated as mean scores and can range from 1 to 7. Higher scores indicate more savoring.
Self-compassion | Change from baseline self-compassion at 3 weeks (T1) and change from baseline mental well-being at 3 months (T2)
  Measured with the 8-item self-reassurance subscale of the Forms of self-criticising/attacking & self-reassuring scale. Scores are calculated as mean scores and can range from 0 to 4. Higher scores indicate more self-compassion.
Positive reframing | Change from baseline positive reframing at 3 weeks (T1) and change from baseline mental well-being at 3 months (T2)
  Measured with 2 items of the positive reframing subscale of the Coping Orientations and Problems Experienced inventory. Scores are calculated as mean scores and can range from 1 to 4. Higher scores indicate more positive reframing.
Anxiety symptoms | Change from baseline anxiety symptoms at 3 weeks (T1) and change from baseline mental well-being at 3 months (T2)
  Measured with the 7-item Generalized Anxiety Disorder-7 questionnaire. Scores are calculated as sum scores and can range from 0 to 21. Higher scores indicate more anxiety symptoms.
Depression symptoms | Change from baseline ability to adapt at 3 weeks (T1) and change from baseline mental well-being at 3 months (T2)
  Measured with the 9-item Patient Health Questionnaire-9. Scores are calculated as sum scores and can range from 0 to 27. Higher scores indicate more depression symptoms.
Spiritual well-being | Change from baseline spiritual well-being at 3 weeks (T1) and change from baseline mental well-being at 3 months (T2)
  Measured with the 7-item Spiritual Attitude and Involvement List-Short Form. Scores are calculated as mean scores and can range from 1 to 6. Higher scores indicate more spiritual well-being.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Twente, Enschede, Overijssel, Netherlands

IPD SHARING:
Plan to Share IPD: Yes